CLINICAL TRIAL: NCT04474587
Title: Impact of Noninvasive Ventilation on Resting Energy Expenditure in Patients With Obesity Hypoventilation Syndrome Treated by Long-term Home Noninvasive Ventilation.
Brief Title: Resting Energy Expenditure in Patients With OHS Treated With Long-term NIV
Status: Suspended | Type: Observational
Why Stopped: COVID pandemic
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Jean-Paul Janssens, University Hospital, Geneva
Other Study IDs: 2020-01223
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Obesity-hypoventilation Syndrome; Resting Energy Expenditure; Long-term Non-invasive Ventilation
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHS-NIV: Patients with obesity-hypoventilation syndrome (OHS) treated with non-invasive ventilation (NIV).
  Interventions: Other: Indirect calorimetry

INTERVENTIONS:
Other: Indirect calorimetry — Measurements of REE by indirect calorimetry

SUMMARY:
This study aims to compare, in subjects with obesity-hypoventilation syndrome (OHS) treated by long-term non-invasive ventilation (NIV), resting energy expenditure (REE) in spontaneous breathing and under NIV. The hypothesise of this study is that REE will be lower under NIV than under spontaneous breathing.

DETAILED DESCRIPTION:
This is an observational monocentric study in which each subject will be its own control. Patients' resting energy expenditure will be measured at rest ("spontaneous breathing" condition) and under its usual treatment ("under NIV" condition) in a cross-over fashion. Conditions measurement order will be randomly generated by a computer algorithm such that half of the patients will be measured under spontaneous breathing before under NIV and the other half of the patients will be measured under NIV before under spontaneous breathing. Resting energy expenditure will be monitored during a short-term elective hospitalization (24 hours). Albeit for measurements of REE, tests which will be performed are part of the regular follow-up of patients under long term NIV.

Primary objective is to compare in OHS patients the REE under spontaneous breathing and under NIV, using their usual settings.

Description of the intended procedures and stages:

1. Recruitment and screening of patients fulfilling inclusion criteria will be done among patients with OHS under long-term NIV followed by our center (duration: 14 days).
2. Once informed written consent has been provided, patients will be included in the study protocol (time provided for decision: 28 days).
3. Patients are admitted for one night with overnight recording of nocturnal oximetry and transcutaneous capnography using their noninvasive ventilation at usual settings, prior to measurements of resting energy expenditure. Downloading of memorized data by ventilator software will also take place and will cover the previous month and the night of the study (duration: 12 hours). These procedures are part of the routine evaluation of patients under long term NIV.
4. Body weight will be measured, as well as body composition by bioelectrical impedance: briefly, a very low intensity electric current is sent between 2 electrodes placed on the dorsum of the foot and the ipsilateral hand. Measurement of resistance and reactance allows estimation of body compartments (fat-free mass and fat mass) (duration: 30 minutes).
5. Patients will undergo their first indirect calorimetric measurement. Prior to REE measurements, patients must be fasting for at least 10 hours, in a supine position, or if required for patient comfort, with a 30° inclination of head rest for at least 30 minutes. REE measurements are either performed with or without noninvasive ventilation (conditions order will be randomized by a computer)(duration: 30 minutes of rest and 20-30 minutes of indirect calorimetry).
6. Interval between measurements of at least 1 hour, to avoid impact of noninvasive ventilation on measurements. Between tests, they will perform pulmonary function tests and have their arterialized capillary blood gases sampled at earlobe (duration: 1 hour). These tests are part of the routine evaluation of patients under long term NIV.
7. Patients will undergo their second indirect calorimetric measurement (see details in section on indirect calorimetric). Prior to REE measurements, patients must be fasting for at least 10 hours, in a supine position, or if required for patient comfort, with a 30° inclination of head rest for at least 30 minutes. REE measurements are either done with or without noninvasive ventilation (randomized order by a software) (duration: 30 minutes of rest and 20-30 minutes of indirect calorimetry).
8. These two tests will be performed in a randomized order (spontaneous breathing or noninvasive ventilation).
9. Information to the patient of the results, which will also be forwarded to physician and nutritionist in charge.

In 2016-2017, seventy-four OHS patients treated at home by long-term NIV were identified in our area. Expecting a participation rate of around 50%, at least 30 patients will be included in the present study. With such a sample size, the study will have a power of 80% to detect an effect size of 0.5.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill all criteria of obesity hypoventilation syndrome.
* Under home NIV for at least 3 months.
* Are compliant to their treatment of NIV (defined as a daily median use > 3:30 hours).
* Have a satisfactory response to NIV (defined by a daytime PaCO2 in a sitting position < 6.5 kPa, and a mean nocturnal SpO2 > 90%, with less than 20% of total recording time spent with an SpO2 < 90%).
* Are in a stable clinical condition (i.e. no episode of acute cardiac and/or respiratory failure leading to a hospitalization within the preceding 3 months).
* Are over 18 years of age.
* Are able to provide informed consent.
* Agree to participate in the study.

Exclusion Criteria:

* Presents any respiratory disorder other than OHS.
* Has been under NIV less than 3 months.
* Is noncompliant (defined above) and/or intolerant to NIV.
* NIV not reaching the above-mentioned physiological targets (defined by a daytime PaCO2 in a sitting position < 6.5 kPa, and a mean nocturnal SpO2 > 90%, with less than 20% of total recording time spent with an SpO2 < 90%).
* Had a recent episode of cardiac and/or respiratory failure leading to a hospitalization within the preceding 3 months.
* Is under 18 years of age.
* Presents a situation interfering with understanding of the protocol and ability to provide informed written consent (language barrier, cognitive disorder, psychiatric disturbance).
* Refuses to participate in the study.
* Is under nocturnal oxygen supplementation on NIV.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with obesity hypoventilation syndrome (OHS) trated with non-invasive ventilation (NIV).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
REE | Each procedure (indirect calorimetry) will take 30 minutes
  Resting energy expenditure (REE) and will be determined under spontaneous breathing and under NIV with an indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland